CLINICAL TRIAL: NCT01059305
Title: Phase II Trial of Erlotinib, a Small Molecule Tyrosine Kinase Inhibitor of EGFR, Prior to Surgery or Radiation in Patients With Aggressive Squamous Cell Cancers (SCC) of the Skin
Brief Title: Phase II Trial of Erlotinib, Prior to Surgery or Radiation in Patients With Squamous Cell Cancers (SCC) of the Skin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of primary outcome efficacy.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0723; NCI-2011-00252 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Skin Cancer
Keywords: Erlotinib; Erlotinib Hydrochloride; OSI-774; Tarceva; Squamous cell carcinoma of the skin; Aggressive cutaneous squamous cell carcinoma; CSCC; Local surgery; Radiation therapy; Epidermal growth factor receptor; EGFR; Small Molecule Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Skin Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib (Experimental): 150 mg daily by mouth before surgery and/or radiation therapy (Induction Treatment); and after surgery and/or radiation erlotinib for up to 1 year (Maintenance Phase).
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — 150 mg daily by mouth before surgery and/or radiation therapy (Induction Treatment); and after surgery and/or radiation erlotinib for up to 1 year (Maintenance Phase).
  Other Names: OSI-774; Erlotinib Hydrochloride; Tarceva

SUMMARY:
The goal of this clinical research study is to learn if Tarceva ® (erlotinib) when taken before and after radiation and/or surgery can help to control aggressive cutaneous squamous cell carcinoma. The safety of the drug will also be studied.

DETAILED DESCRIPTION:
Erlotinib is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Study Treatment/Study Drug Administration:

If you are found to be eligible to take part in this study, you will take erlotinib before surgery and/or radiation therapy (Induction Treatment). After surgery and/or radiation you will take erlotinib for up to 1 year (Maintenance Phase).

Induction Treatment:

You will take erlotinib 1 time every day, by mouth, with a full glass of water.

You will take erlotinib at about the same time every day. If you miss a dose and there is at least 12 hours before the next dose is due, you will need to take the missed dose. You should then take your next dose as scheduled. If you vomit after taking the tablet, the dose should be replaced only if the tablet can actually be seen. Erlotinib should be taken 1 hour before and 2 hours after meals and other drugs.

If you have side effects from erlotinib, the study doctor may lower your dose.

When you stop taking erlotinib during induction will depend on if the disease gets worse, if the doctor thinks you are benefitting, and if you will receive surgery and/or radiation.

You will take erlotinib for up to 10 weeks before starting local therapy. If the doctor thinks you are benefitting, you may take erlotinib for longer than 10 weeks before starting surgery and/or radiation. If the disease gets worse before 10 weeks, you will stop taking erlotinib and have surgery and/or radiation right away.

Surgery/Radiation:

During Week 4, the doctor will decide if the disease is resectable or unresectable and will schedule the type of local therapy (surgery and/or radiation) that you will receive. If You will sign separate consents for the surgery and/or radiation, which will describe the procedure(s) and the risks in detail.

Resectable Disease:

If the disease is resectable, you will be scheduled to have surgery. If the doctor thinks it is needed, you may have radiation therapy after the surgery. Radiation therapy usually will start 4-8 weeks following your surgery, if the surgical site has healed.

You will take erlotinib until 7 days before your surgery.

Unresectable Disease:

If the disease is unresectable, you will be scheduled to have radiation therapy.

You will take erlotinib until you begin the radiation therapy. If your doctor thinks you are benefiting from erlotinib, you will continue taking it during the radiation therapy.

After you complete your radiation therapy, if the doctor thinks it is needed, you will have surgery.

Maintenance Treatment:

You will restart erlotinib at 4-8 weeks after surgery, if the surgical site has healed. If you have radiation therapy after the surgery, you will take erlotinib during the radiation treatment.

If you only received radiation therapy, you will continue erlotinib after you finish your radiation therapy.

You will take erlotinib by mouth every day for up to 1 year.

Study Visits:

Induction Therapy:

On Day 1 before Induction Therapy and then every 2 weeks:

* You will be asked be asked about any side effects you may have had and any drugs you may be taking.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about your smoking status.
* Your performance status will be recorded.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* The tumor will be measured by physical exam using rulers and/or calipers.
* Pictures will be taken of the same areas that were photographed during screening.
* If you are taking anti-coagulant medication, blood (about 1-2 teaspoons) will be drawn to check your blood clotting function.
* If your doctor thinks it is needed, you will have an ECG.

After Week 4, you will have a CT scan or MRI scan to check the status of the disease. If you continue taking erlotinib for at least 4 more weeks (a total of 8 weeks) before surgery or radiation is started, the CT or MRI will be repeated then.

After Week 4 and within 14 days before you start maintenance therapy, you will complete questionnaires about how you are feeling and your overall quality of life. The questionnaires will take about 10-15 minutes total to complete.

Maintenance Therapy:

On Day 1 before Maintenance Therapy and then every 8 weeks:

* You will be asked about any side effects you have had and any drugs you may be taking.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about your smoking status.
* Your performance status will be recorded.
* The tumor will be measured.
* Pictures will be taken of the same areas that were photographed during screening.
* If the doctor thinks it is needed, you will have a CT scan or MRI scan to check the status of the disease.
* If your doctor thinks it is needed, you will have an ECG
* Blood (about 2-3 teaspoons) will be drawn for routine tests, including tests to check your blood clotting function (Day 1 only).
* If you are taking anti-coagulant medication, blood (about 2-3 teaspoons) will be drawn to check for blood clotting function (every 8 weeks only).

After Weeks 24 and 52, you will complete the questionnaires about how you are feeling and your overall quality of life.

If you only received radiation therapy, you will have a CT scan or MRI scan 3 months after the radiation therapy.

Length of Study:

You will take the study drug for up to 1 year after the surgery/radiation. You will be taken off study if the disease gets worse, if you have intolerable side effects, or if the doctor thinks it is in your best interest to stop.

End-of-Treatment Visit:

About 30 days after the last dose of study drug, the following tests and procedures will be performed:

* You will be asked about any side effects you may have had and about any drugs you may be taking.
* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a CT scan or MRI to check the status of the disease.

Long-Term Follow-Up:

After the end-of-treatment visit, you will be contacted every 3 months during Year 1 and every 6 months during Years 2 and 3 to collect information about how you are doing, any treatment you have received, and any other side effects you have experienced. You (or your family members or designees) may be contacted by telephone, in writing, by e-mail, or during clinic visits. This information may also be collected by checking your medical record. This follow-up will also consist of a physical exam if you are being seen at MD Anderson for your follow-up.

This is an investigational study. Erlotinib is FDA approved and commercially available for the treatment of non-small cell lung cancer. It is investigational to give erlotinib before and after radiation and/or surgery for the treatment of aggressive cutaneous squamous cell carcinoma.

Up to 25 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Within 12 weeks prior to study entry, patient must have histologically or cytologically confirmed cutaneous squamous cell carcinoma (CSCC) that is either locally advanced or recurrent, and no evidence of distant metastases. If the biopsy was collected outside of MD Anderson Cancer Center (MDACC), the MDACC Pathology Department must assess and confirm the SCC diagnosis.
2. Patient is eligible with previous surgical intervention if they have residual or recurrent disease, it is greater than 6 weeks since surgery and they have fully recovered from the surgery.
3. Patient must have measurable disease.
4. Tumor must be at least 2 centimeters in size as measured by the treating physician(s) or PI, or have histological or cytological verification of muscle, bone, lymph node metastasis, or perineural involvement,.
5. Surgical resection or radiation must be planned as part of the treatment strategy for the CSCC.
6. At least 18 years of age.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
8. Must have adequate organ and marrow function as follows:(a) leukocytes >/= 3,000/mm^3 (b) absolute neutrophil count >/= 1,500/mm^3 (c) platelets >/= 75,000/mm^3 (d) hemoglobin >/= 8g/dL (e) total bilirubin </= 2 X institutional upper limit of normal (ULN) (f) AST(SGOT)/ALT(SGPT) </= 2.5 X ULN if alkaline phosphatase is normal, or alkaline phosphatase </= 4 x ULN if transaminases are normal (g) Creatinine </= 2.0 x ULN or creatinine clearance >/= 60 mL/min/1.73 m^2
9. Must be able to take intact tablets by mouth, or be able to take tablets dissolved in water by mouth or by a percutaneous gastrostomy tube.
10. Patients - both males and females - with reproductive potential (includes women who are menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Birth control should continue for 4 weeks after discontinuation of erlotinib therapy. Women of childbearing potential must provide a negative pregnancy test (serum betaHCG) within within 72 hours prior to first receiving protocol therapy.
11. Must have ability to understand and the willingness to sign a written Informed Consent Document (ICD). In the event that non-English speaking participants are eligible for this study, a short form (if applicable) or an ICD in their language will be utilized and completed in accordance with the MDACC "Policy For Consenting Non-English Speaking Participants."
12. Must be willing to receive their definitive local therapy, that is surgery and / or radiation therapy, at M. D. Anderson Cancer Center.
13. Organ transplant patients are eligible as long as they do not have active signs of rejection and have adequate bone marrow function.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or have child-bearing potential & are unwilling/unable to use an acceptable method of contraception for the entire study period & for at least 4 weeks after cessation of the study drugs. If the pregnancy test is positive, the patient must not receive erlotinib, & must not be enrolled on the study. Erlotinib is a signal transduction inhibitor agent w/ the potential for teratogenic or abortifacient effects.
2. -continued from Exclusion #1- If the pregnancy test is positive, the patient must not receive erlotinib, and must not be enrolled on the study. Erlotinib is a signal transduction inhibitor agent with the potential for teratogenic or abortifacient effects. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with erlotinib, breastfeeding should be discontinued if the mother is treated with erlotinib.
3. Patient with distant metastatic disease.
4. Patient who has had previous radiotherapy to the site of the skin cancer being treated on this protocol.
5. Patient currently receiving any other anticancer or investigational agents at time of study enrollment.
6. Patient has received prior EGFR inhibitor therapy.
7. Patient with a history of an invasive malignancy (other than the one treated in this study) or lymphoproliferative disorder within the past 5 years. Patients with a history of adequately treated non-melanoma skin cancer, ductal carcinoma in situ of the breast or carcinoma in situ of the cervix are allowed.
8. Patient with history of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib.
9. Patient is unwilling or unable to discontinue prohibited concomitant therapies.
10. In the opinion of the investigator, patient with any condition that is unstable or could jeopardize the safety of the patient or could limit compliance with the study's requirements. These include, but are not limited to, ongoing or active infection requiring parenteral antibiotics at time of study registration, psychiatric illness that would limit compliance with study requirements or symptomatic congestive heart failure (NYHA class II or greater), unstable angina pectoris or cardiac arrhythmia requiring maintenance medication.
11. Patient with a history of pulmonary fibrosis (other than in a radiated field) or chronic liver disease.
12. Patients with active gastrointestinal disease or a disorder that alters gastrointestinal motility or absorption; for example, a significant surgical resection of the stomach or small bowel, uncontrolled inflammatory bowel disease or uncontrolled chronic diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S. Glisson, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Process: February 15, 2011 to September 11, 2012. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Erlotinib: 150 mg daily orally before surgery and/or radiation therapy (Induction Treatment); and after surgery and/or radiation erlotinib for up to 1 year (Maintenance Phase).
Period: Overall Study
Arm/Group | Erlotinib
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 70 [58 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Response Evaluation Criteria In Solid Tumors (RECIST) criteria for CR = complete response, PR = partial response, SD = stable disease, PD = progressive disease, and NE = inevaluable. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): >30% decrease in sum of diameters of target lesions, reference baseline sum diameters. Progressive Disease (PD): >20% increase in sum of diameters of target lesions, reference smallest sum on study (this includes baseline sum if is smallest on study). In addition to relative increase of 20%, sum must absolute increase at least 5 mm. (Note: appearance of 1/> new lesions also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum diameters while on study. Not evaluable (NE): Inevaluable when no imaging/measurement done
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 10
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 7
  Progressive Disease | 2

ADVERSE EVENTS:
Time Frame: Adverse events collected through maximum of 10 weeks of Erlotinib treatment.
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Cholesterol high (Investigations) | 3 (3)
Concentration impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (8)
Dizziness (Nervous system disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Eye pain (Eye disorders) | 2 (2)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Dental Infection (Infections and infestations) | 1 (1)
INR increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Paronychia (Infections and infestations) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 (7)
Skin infection (Infections and infestations) | 1 (2)
Stroke (Nervous system disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes